CLINICAL TRIAL: NCT07350720
Title: Inpatient Care of Patients With Difficult to Treat Eating Disorders - What Affects Treatment Outcome?
Brief Title: Inpatient Care of Patients With Difficult to Treat Anorexia Nervosa - Factors Affecting Treatment Outcome.
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-07313-01
Record Dates: First submitted 2025-12-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorders; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of the project is to investigate factors that may influence treatment outcomes in people with difficult-to-treat anorexia nervosa who are enrolled in inpatient care at the Region Skåne Eating Disorders Centre in Lund. Treatment expectations, sense of autonomy, and patient participation, will be investigated, as well as caregivers' attitudes towards, and experiences of working with, autonomy and patient participation in the inpatient setting. The research project is expected to contribute to increased knowledge about the treatment of difficult-to-treat anorexia nervosa, and what part patient participation and autonomy may play when treating severe eating disorders. The overall objectives of the research program are:

1. To contribute to increased knowledge about factors that influence the treatment of people with difficult-to-treat anorexia nervosa
2. To highlight the role of autonomy and patient participation in inpatient care of severe eating disorders
3. To use the research results for clinical improvement work at Region Skåne Eating Disorders Center

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa diagnosis (ICD F50.0)
* Admitted to inpatient care at department 5 at Region Skåne Eating Disorders Center

Exclusion Criteria:

* Confidential identity
* Inability to read or write in Swedish or English
* Condition or treatment that, according to the study team, makes participation in the study inappropriate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with anorexia nervosa admitted to inpatient care at Region Skåne Eating Disorders Center, a specialized psychiatric care unit for treatment of eating disorders.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | BMI will be calulated on a weekly basis throughout the inpatient treatment period, and baseline measures until end of treatment/discharge from inpatient unit at approximately 12 weeks will be used for analysis.
  BMI is calculated using weight and height: weight (kg) / (height (m) x height (m))

SECONDARY OUTCOMES:
Treatment satisfaction | CSQ-8 is collected at the end of treatment/at discharge from inpatient care at approximately 12 weeks as well at 1 year follow-up after discharge, in order to evaluate the treatment given.
  Satisfaction with treatment will be measured using the Client Satisfaction Questionnaire (CSQ-8), which contains 8 items. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Emelia Mellergård, PhD, Principal Investigator — Region Skåne VO Vuxenpsykiatri Lund

IPD SHARING:
Plan to Share IPD: No